CLINICAL TRIAL: NCT03651284
Title: Project LiGHT (Living Green and Healthy for Teens): A Novel Weight Management Program That Emphasizes the Benefits of a Healthy Lifestyle
Brief Title: Investigating the Efficacy of a Mobile App Intervention to Change Youth and Their Families' Health Behaviours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Childhood Obesity Foundation (Other); Ayogo Health Inc. (Other); Public Health Agency of Canada (PHAC) (Other Government); Merck Canada Inc. (Industry); Pacific Blue Cross (Unknown); Heart and Stroke Foundation of Canada (Other); David Suzuki Foundation (Unknown); Craving Change (Unknown); Diabetes Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government); British Columbia Children's Hospital (Other); Children's Hospital of Eastern Ontario Research Institute (Other); The Hospital for Sick Children (Other); Hamilton Health Sciences Corporation (Other); Alberta Health services (Other); The Governors of the University of Alberta (Unknown); University of Alberta (Other); Alberta Innovates Health Solutions (Other); Women and Children's Health Research Institute, Canada (Other); Canadian Obesity Network (Unknown); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Louise Masse, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H16-03090-b
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Obesity, Pediatric
Keywords: obesity; physical activity; nutrition; adolescents; gamification; video game; sedentary activity
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim2Be Live Coach (Experimental): Aim2Be app with Live Coach + Fitbit + BMI tracking tools
  Interventions: Behavioral: Aim2Be app with Live Coach + Fitbit + BMI tracking tools
- Aim2Be Waitlist (Other): Aim2Be app waitlist + Canadian Health Recommendations + Fitbit + BMI tracking tools for three months, then flip to Aim2Be app with Virtual Coach + Fitbit + BMI tracking tools
  Interventions: Behavioral: Aim2Be app waitlist + Canadian Health Recommendations + Fitbit + BMI tracking tools, then flip to Aim2Be app with Virtual Coach + Fitbit + BMI tracking tools

INTERVENTIONS:
Behavioral: Aim2Be app with Live Coach + Fitbit + BMI tracking tools — Participants will spend six months using the Aim2Be app setting aims, completing tasks, accessing articles, doing self-assessments, and participating in the social wall. They will also complete a series of questionnaires, dietary recalls, BMI tracking using scales and tape measures, and physical activity tracking using Fitbits. Participants in this condition will have access to the Live Coach and the Virtual Coach. The Live Coach has specialized training in lifestyle and motivational interviewing and will support families in changing their health behaviours through in-app messaging and phone calls. The Virtual Coach gives guidance to families through an avatar that has been programmed using motivational interviewing theory.
  Arms: Aim2Be Live Coach
Behavioral: Aim2Be app waitlist + Canadian Health Recommendations + Fitbit + BMI tracking tools, then flip to Aim2Be app with Virtual Coach + Fitbit + BMI tracking tools — Participants in this condition will be waitlisted for three months while they receive standard of care (Canadian Health Recommendations for physical activity, dietary habits, screen behaviours, and sleep). Participants will gain access to the Aim2Be app with Virtual Coach after the three month assessment. Participants will then spend three months using the Aim2Be app setting aims, completing tasks, accessing articles, doing self-assessments, and participating in the social wall. For the whole six months, participants will complete a series of questionnaires, dietary recalls, BMI tracking using scales and tape measures, and physical activity tracking using Fitbits. Participants in this condition will have access to the Virtual Coach only. The Virtual Coach gives guidance to families through an avatar that has been programmed using motivational interviewing theory.
  Arms: Aim2Be Waitlist

SUMMARY:
This study is the second of three sub-studies aimed at evaluating the outcomes of the Living Green and Healthy for Teens (LiGHT) program, delivered through the Aim2Be app (v2.2). Aim2Be is an app for 10 to 17 year olds and their families that is intended to help them shift from an healthy lifestyle toward better health habits in four areas: nutrition, physical activity, recreational screen time, and sleep. This second evaluation has the following aims to: 1) describe reach; 2) assess change in knowledge of Canadian health recommendations; and 3) assess change in lifestyle behaviours and weight outcomes and whether these changes are moderated by involvement in the app. This study uses a two-group parallel/crossover randomized controlled trial design following N=200 families for six months.

DETAILED DESCRIPTION:
Living Green and Healthy for Teens (LiGHT v2) is an engaging online, individualized, gamified lifestyle management program for youth, delivered through the Aim2Be app. LiGHT v2 is focused on initiating long-term behaviour change in youth and their families in order to help them shift from an unhealthy lifestyle toward better health habits in four areas: nutrition, physical activity, recreational screen time, and sleep. The program aims to support healthy lifestyles of 10- to 17-year-old children and adolescents, as well as to mitigate increased risk for metabolic and non-metabolic complications associated with obesity in the short and long term.

The app includes content that involve the family, and focus on behavioural therapy as well as dietary and physical activity patterns. Aim2Be is intended to be engaging and fun, provide virtual and tangible rewards, interact with participants multiple times per day, and provide a mobile social support network.

Pre-teens (10-13) and teens (14-17) will each have their own unique versions of Aim2Be. Content will be tailored specifically to the developmental stage and needs of each age group. The content will be delivered in such a way that it facilitates education, peer-to-peer conversation, and self-regulation in an engaging platform.

Because parents have been shown to be of primary importance in supporting healthy lifestyles of children, LiGHT v2 will educated and engage parents as well as youth. Parents will receive separate, but complementary content, intended to guide them as they shop for and prepare food and make behavioural changes within their families. The content for parents will be delivered using the same social aspects of Aim2Be as the pre-teens and teens, but the channels will be gated, so teens and parents each have their own space. Aim2Be's social features will help parents strategize and empathize with other families who wish to adopt healthy lifestyles.

The program will be evaluated using three separate study groups. This protocol describes the second of the three.

Families (one parent and one child) will be recruited through advertising on social media and through active referral from six Canadian Pediatric Weight Management Registry (CANPWR) sites (Children's Hospital of Eastern Ontario, SickKids, McMaster Children's Hospital, Stollery Children's Hospital, Alberta Children's Hospital, and British Columbia Children's Hospital). Approximately 350 families will be recruited and a total of 200 families will be enrolled into the study and randomized into two groups. This study uses a two-group parallel/crossover randomized controlled trial design. All families will be given access to Aim2Be v2.2 to use from their mobile device or home computer. Participants will be prospectively followed for six months.

Once participants are deemed eligible to participate in the study and complete their baseline assessments, they are allocated to one of two conditions: 1) Live Coach; or 3) waitlist control group given standard of care. Participants in the Live Coach group will be given access to Aim2Be for six months with a live coach who has expertise in supporting lifestyle modification and will help youth and parents set goals and achieve these goals using principles from motivational interviewing. Participants in the control group will be wait listed for enrollment in the app for three months and will be given access to the Virtual Coach version of the app after they complete the three month evaluation. The Virtual Coach group version provides automated guidance from a virtual coach instead of a live person, but that is programmed using the same motivational interviewing principles.

Evaluation at baseline, three months, and six months will be used to compare whether those assigned to the different coach conditions have better health outcomes than those assigned to the waitlist control group. Parents will complete questionnaires at baseline, three months, and six months, which assess sociodemographics, behaviours, and mediators of behaviour change. Youth will complete questionnaires at baseline, three months, and six months, which assess health behaviours, mediators of behaviour change, and knowledge of Canadian recommendations for healthy behaviours. Questionnaire data will be collected and managed using REDCap.

Families will be provided with a Fitbit, scale, and measuring tape when they enroll in the study. At each assessment point (baseline, three months, and six months), parents will provide youth's height and weight, and youth will complete three 24-hour dietary recalls and wear the Fitbit for the duration of the study.

Honoraria will be paid at each time point to compensate participation.

Participants will be randomly allocated to each of the two groups and have equal likelihood of assignment to each condition. Participants will not be blinded as the design of the intervention does not facilitate this. Participants will be informed of their allocation after completing all baseline measures. Evaluators and researchers will be blinded to allocation during data analysis.

The aims of this study are to: 1) determine reach/ who participates in this study (short term outcome); 2) determine whether participation in the program increases adolescents' knowledge of Canadian health recommendations related to dietary habits, physical activity, and sedentary behaviour (medium term outcome); and 3) assess the impact of Aim2Be on changes in dietary habits, physical activity, and sedentary behaviours as well as Body Mass Index (BMI) and whether the impact is moderated by involvement in the app (long term outcome).

ELIGIBILITY:
Inclusion Criteria:

* Child must be between 10 and 17 years old
* Child and at least one of their parents must be able to read at the grade 5 level or above
* Parent participant must be the caregiver with whom the child primarily lives
* Families must have a computer or mobile device and internet access at home
* Child participants must be either overweight or obese, as defined by the age and gender specific WHO cut-offs for children and adolescents aged 5 to 19

Exclusion Criteria:

* Diagnosis of any musculoskeletal, cardiovascular, pulmonary, or orthopedic problems or disabilities precluding the participant from being physically active
* Any other physical condition that precludes the participant from being physically active
* Diagnosis of anorexia nervosa or bulimia nervosa
* Diagnosis of Type I diabetes
* Dietary restrictions or special diets that limit a participant's ability to eat a variety of foods
* Simultaneous participation in another physical activity, nutrition, or weight management study/program
* Use of medication, nutritional supplements, or herbal preparations to help lose weight
* Pregnancy
* A history of psychiatric problems or substance abuse which would interfere with adherence to the study protocol

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index z-score (youth) | Baseline, 3 months, 6 months
  Change in BMI z-scores will be computed from measured height and weight using World Health Organization (WHO) cut-offs
Change in health behaviour knowledge (youth) | Baseline, 3 months, 6 months
  Survey questions (using a LiGHT-specific tool) will assess teens' knowledge of Canadian recommendations for healthy eating, physical activity, and sedentary behaviours. Knowledge will be reported as an aggregate knowledge score from 0 to 8 (a score of 0 indicates low knowledge and a score of 8 indicates high knowledge), as well as sub-score for each of the knowledge areas (nutrition, physical activity, recreational screen time, sleep).
Change in objective dietary behaviour (youth) | Baseline, 3 months, 6 months
  Change in mean daily servings of fruits and vegetables and sugar-sweetened beverages consumed over three consecutive 24-hour dietary recalls.
Change in number of daily steps (youth) | Baseline, 3 months, 6 months
  Change in mean daily steps over a 14-day period at each assessment point, as measured using a Fitbit activity monitor.
Change in screen behaviour (youth) | Baseline, 3 months, 6 months
  Survey questions will assess adolescents' recreational screen time use (using the Take Action survey), and will be reported as the number of self-reported hours of recreational screen time per day.

SECONDARY OUTCOMES:
Adherence | 3 months, 6 months
  App analytics will be used assess participants' adherence to the intervention
Reach | Baseline
  Survey questions will assess socio-demographic characteristics of families and will be compared against families who typically register for weight-management centres in Canada.
Change in Healthy Eating Index score (youth) | Baseline, 3 months, 6 months
  Change in score of dietary quality, as measured using three consecutive 24-hour dietary recalls and scored on the Healthy Eating Index (adapted for the Canadian recommendations).
  Total score: [0-100] (sum of all subscale scores; high scores represent better outcomes)
  Adequacy (high score=high consumption) Total fruits: [0-5] Whole fruits: [0-5] Total vegetables: [0-5] Greens and beans: [0-5] Whole grains: [0-10] Dairy: [0-10] Total protein foods: [0-5] Seafood and plant proteins: [0-5] Fatty acids: [0-10]
  Moderation (high score=low consumption) Refined grains: [0-10] Sodium: [0-10] Added sugars: [0-10] Saturated fats: [0-10]
Change in self-reported dietary behaviour (youth) | Baseline, 3 months, 6 months
  Survey questions will assess adolescents' dietary behaviours, and be reported as average number of servings of fruits and vegetables and consumption of sugar-sweetened beverages per day.
Change in self-reported physical activity behaviour (youth) | Baseline, 3 months, 6 months
  Survey questions will assess adolescents' physical activity behaviours, and change in physical activity will be reported as average number of days they were active for at least 60 minutes. Adolescent physical activity will be assessed using a modified version of the International Physical Activity and the Environment Network Adolescent Survey for Children.
Change in self-reported dietary behaviour (parents) | Baseline, 3 months, 6 months
  Survey questions will assess parents' dietary behaviours, and be reported as average number of fruits and vegetables and sugar-sweetened beverages per day.
Change in self-reported physical activity behaviour (parents) | Baseline, 3 months, 6 months
  Survey questions will assess parents' physical activity behaviours, and change in physical activity will be computed based on a composite physical activity score. Parent physical activity will be assessed using a modified version of the International Physical activity Questionnaire Short Form (IPAQ-SF), and scored as average minutes per day of moderate and vigorous physical activity.
Change in screen behaviour (parents) | Baseline, 3 months, 6 months
  Survey questions will assess parents' recreational screen time use (using the Take Action survey), and will be reported as the number of self-reported hours of recreational screen time per day.
Change in mediators of behaviour change | Baseline, 3 months, 6 months
  Survey questions will assess adolescents' self-efficacy and motivation in changing the health behaviours targeted by LiGHT.

OTHER OUTCOMES:
Functionality | 3 months, 6 months
  Survey questions will assess whether users like the program (i.e. was Aim2Be fun, easy to use and intuitive, did it offer content to which they could relate and features they like).

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Masse, PhD, Principal Investigator — University of British Columbia, BC Children's Hospital Research Institute
Locations (6):
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Tugault-Lafleur CN, De-Jongh Gonzalez O, Macdonald J, Bradbury J, Warshawski T, Ball GDC, Morrison K, Ho J, Hamilton J, Buchholz A, Masse L. Efficacy of the Aim2Be Intervention in Changing Lifestyle Behaviors Among Adolescents With Overweight and Obesity: Randomized Controlled Trial. J Med Internet Res. 2023 Apr 25;25:e38545. doi: 10.2196/38545. PMID 37097726
- [Derived] Deslippe AL, Gonzalez OD, Buckler EJ, Ball GDC, Ho J, Bucholz A, Morrison KM, Masse LC. Do Individual Characteristics and Social Support Increase Children's Use of an MHealth Intervention? Findings from the Evaluation of a Behavior Change MHealth App, Aim2Be. Child Obes. 2023 Oct;19(7):435-442. doi: 10.1089/chi.2022.0055. Epub 2022 Dec 22. PMID 36576875
- [Derived] De-Jongh Gonzalez O, Tugault-Lafleur CN, Buckler EJ, Hamilton J, Ho J, Buchholz A, Morrison KM, Ball GD, Masse LC. The Aim2Be mHealth Intervention for Children With Overweight or Obesity and Their Parents: Person-Centered Analyses to Uncover Digital Phenotypes. J Med Internet Res. 2022 Jun 22;24(6):e35285. doi: 10.2196/35285. PMID 35731547
- [Derived] Masse LC, Vlaar J, Macdonald J, Bradbury J, Warshawski T, Buckler EJ, Hamilton J, Ho J, Buchholz A, Morrison KM, Ball GDC. Aim2Be mHealth intervention for children with overweight and obesity: study protocol for a randomized controlled trial. Trials. 2020 Feb 3;21(1):132. doi: 10.1186/s13063-020-4080-2. PMID 32014057